CLINICAL TRIAL: NCT06977217
Title: Factors Associated With Response to Cardiac Resynchronization Therapy in Heart Failure Patients With Non-LBBB ECG Pattern
Acronym: FACT-CRT
Status: Active, not recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Valentina Kutyifa, Professor of Medicine (Cardiology), Tenured, University of Rochester
Other Study IDs: STUDY00006153
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cardiomyopathies; Heart Failure; Non-left Bundle Branch Block; Cardiac Resynchronization Therapy
Keywords: Cardiomyopathies; Heart Failure; Non-left bundle branch block; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Cardiomyopathies; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CRT-D implantation — Cardiac resynchronization therapy with a defibrillator (CRT-D). This combination device uses a pacemaker and an implantable cardioverter-defibrillator (ICD). It may be recommended for people with heart failure who also have a risk of sudden cardiac death. It can find dangerous heart rhythms and correct them. It can pace the heartbeat or shock the heart out of a dangerous heart rhythm.

SUMMARY:
Cardiac resynchronization therapy with a defibrillator (CRT-D) in heart failure (HF) patients without left bundle branch block (non-LBBB) has been less beneficial to improve outcomes despite being a guideline indicated therapy, posing a significant treatment challenge. However, non-LBBB patients with echocardiography response to CRT-D have better outcomes, and pre-implant variables could predict response, identifying patients who benefit the most. In this study, we plan to enroll 270 HF patients with non-LBBB and guideline-indicated CRT-D implantation to validate our prior echocardiography predictor score, and to identify novel ECG and echocardiography predictors using conventional statistics and machine learning analysis. We will also assess the applicability of such a score for clinical outcomes of HF, ventricular arrhythmias, or death.

DETAILED DESCRIPTION:
Morbidity, mortality, and health care costs of the treatment of systolic heart failure (HF) are rapidly increasing. Cardiac resynchronization therapy with a defibrillator (CRT-D) is cost-effectively reducing HF events and death in HF patients with a wide QRS and low ejection fraction. However, response to CRT-D is not unequivocally present in all patients, with less benefit in those without the presence of an ECG abnormality, left bundle branch block (non-LBBB), posing a significant treatment challenge.

Because of the conflicting and limited data on response to CRT-D in this cohort, it is possible that we currently treat a large proportion of HF patients with non-LBBB who have limited or no benefit from the device. Therefore, better selection of patients for this expensive therapy is warranted. One of our recent studies suggested a clinical benefit in patients with non-LBBB and marked echocardiography response, and identified predictors. However, there is a need to prospectively validate these predictors of echocardiography response to CRT-D in non-LBBB in this hard-to-treat patient population, and identify potential novel ECG and echocardiography predictors, utilizing novel statistical methods of machine learning. We propose a prospective, observational, single-arm study in a currently guideline-indicated cohort to validate and identify predictors of echocardiography response to CRT-D, including novel ECG and echocardiography markers, and to assess subsequent clinical outcomes in 270 HF patients with an implanted CRT-D and non-LBBB ECG pattern.

The primary aim of the study is to prospectively validating our previously identified clinical predictors of echocardiography response to CRT-D in HF patients with non-LBBB that could enable better patient selection.

Our secondary aim is to identify the incremental value of novel ECG and echocardiography variables to predict echocardiography response to CRT-D in non-LBBB patients, including ECG variables of sum absolute QRST integral and ventricular electrical activation delay, and echocardiography-derived variables of left ventricular dyssynchrony and contractility. Then we will apply the developed predictive model to prospectively identify non-LBBB patients with CRT-D at a risk of heart failure, ventricular arrhythmias, or death. Tertiary aim is to identify novel ECG and echocardiography predictors of response in non-LBBB using machine learning analysis.

Study population will include 270 HF patients with non-LBBB and an implanted CRT-D with 6 months echocardiography follow-up analyzed by an echocardiography core lab, and assessing clinical outcomes of heart failure, ventricular arrhythmias, or death.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older (no upper limit)
* Optimal medical therapy for heart failure as established by current guidelines;
* Class IIa or IIb guideline-based indication for CRT-D in non-LBBB patients, including one of the following:
* New York Heart Association (NYHA) class II HF symptoms, LVEF ≤ 30% and QRS≥ 150 ms (IIb);
* NYHA class III-IVa HF, LVEF ≤ 35%, and QRS duration ≥ 150 ms (IIa);
* NYHA class III-IVa HF, LVEF ≤ 35%, and QRS duration 120- 149 ms (IIb)
* Successful CRT-D generator implant

Exclusion Criteria:

* Unable to obtain imaging data from echocardiogram within 1 year prior to CRT-D implant
* Unable to obtain the 20-minute ECG prior to CRT-D implant
* Unable to enroll within 14 days following successful CRT-D generator implant
* Unable or unwilling to follow the study protocol
* Less than 24 months life expectancy at enrollment
* Pregnancy or planned pregnancy in the next 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include 270 HF patients with non-LBBB and an implanted CRT-D device.
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
LVESV improvement | 12 months
  The primary endpoint of the study is a 25% or greater reduction in LV end-systolic volume 12 months after CRT-D implantation in HF patients with non-LBBB, analyzed by the central echocardiography core laboratory. Echocardiography outcomes will be assessed by sonographers blinded to patient characteristics or clinical outcomes to avoid bias.

SECONDARY OUTCOMES:
HF or death or VT or VF | 2 years
  Secondary endpoints will include the composite of heart failure, death, and device detected ventricular tachycardia or ventricular fibrillation to account for all types of adverse outcomes in HF patients with CRT-D.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Kutyifa, MD, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States